CLINICAL TRIAL: NCT04021888
Title: The Effects of Exercise Program in Alzheimer's Patients With Mild to Moderate Stage Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dokuz Eylul University (Other)
Collaborators: Sevgi Ozalevli (Unknown); Gorsev Yener (Unknown)
Responsible Party: Principal Investigator, Elvan Keles, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KELES
Record Dates: First submitted 2019-07-13; First posted 2019-07-16 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Alzheimer Disease; Aerobic Exercise; Breathing Exercise; Resistance Training
MeSH Terms: conditions — Alzheimer Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An assessor who was blinded to treatment groups assessed clinical outcomes before the treatment process. The same assessor was also repeated assessments at 13th week (at the end of treatment process)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental)
  Interventions: Other: Exercise
- Control (Active Comparator)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Education of patients and their caregivers, deep breathing exercise, aerobic exercise and resistance training with elastic bands

SUMMARY:
The primary aim of this trial is to investigate the feasibility of an exercise program consisting of respiratory exercises, aerobic exercises and strengthening exercises in mild to moderate Alzheimer's disease. The trial also aims to investigate the effectiveness of the exercise program on respiratory symptoms, exercise capacity, cognition, physical performance, depression, sleepiness, activities of daily living and quality of life.

Patients will be divided into exercise (intervention) and control group by randomization method. The study is planned to be performed with a total of 60 patients, 30 in each group. The patients in the exercise group will be given breathing exercises aerobic exercises and strengthening exercises for 2 days a week for 12 weeks, about 30-40 minutes while the patients in the control group will be provided with suggestions, home exercise program and daily life activities

DETAILED DESCRIPTION:
Exercise group was trained 3 times a week under the supervision of a physiotherapist and encouraged to exercise at home on other days

ELIGIBILITY:
Inclusion Criteria:

* aged over 65 years
* can walk independent

Exclusion Criteria:

* can't see
* have done any exercise in the last 6 months
* have a major and uncontrolled orthopedic, neurological or cardiopulmonary problem that restricts functioning
* having non Alzheimer's disease dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in cognition | Baseline, 12th week
  The Mini-Mental State Examination (MMSE) is used to measure cognitive impairment in older adults. It assesses different subset of cognitive status including attention, language, memory, orientation, visuospatial proficiency.

SECONDARY OUTCOMES:
Change in pulmonary functions | Baseline, 12th week
  Pulmonary function test (PFT) is a generic term used to indicate a battery of studies or maneuvers that may be performed using standardized equipment to measure lung function.
Change in respiratory muscle strength | Baseline, 12th week
  Measurement of respiratory muscle strength is useful in order to detect respiratory muscle weakness and to quantify its severity. Respiratory muscle strength is assessed by mouth pressures sustained for 1 s during maximal static manoeuvre against a closed shutter
Change in functional capacity | Baseline, 12th week
  Six-minute walk test (6MWT) is a valid, reliable and useful test for assessing functional capacity of COPD patients. This test assesses distance walked over 6 minutes as a sub maximal test of aerobic capacity/endurance.
Change in physical performance | Baseline, 12th week
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people.
Change in sleepiness | Baseline, 12th week
  The Epworth sleepiness scale (ESS) is a questionnaire that's routinely used to assess daytime sleepiness. The person filling in the questionnaire rates how likely they are to doze off during the day in different situations.
  Patients scored eight questions according to the probability of sleeping 0, 1, 2, 3, and the sum of the eight questions was calculated. A high score indicates sleepiness. If the total score is greater than 10, it indicates the presence of pathological sleepiness.
Change in quality of life | Baseline, 12th week
  The Alzheimer's Disease-Related Quality of Life (ADRQL), is consist of 13-item self-report and 13- item caregiver-report measures. Each item is evaluated on a 4-point scale (1 point is bad and 4 points is excellent)
Change in activities of daily living | Baseline, 12th week
  Barthel Index for Activities of Daily Living (ADL) measures functional disability by quantifying patient performance in 10 activities of daily life. These activities can be grouped according to self-care (feeding, grooming, bathing, dressing, bowel and bladder care, and toilet use) and mobility (ambulation, transfers, and stair climbing). Points are given according to doing daily life activities dependently or independently. It ranges from 0 to 100 and 0 points refers to complete dependence, 100 points refers to independence The Lawton Instrumental Activities of Daily Living (IADL) Scale assesses a person's ability to perform tasks such as using a telephone, doing laundry, and handling finance. This scale consist of 8 question. Higher values represent a better outcome.
Change in depression | Baseline, 12th week
  The Geriatric Depression Scale-Short Form (GDS-SF) is an instrument that was developed to assess depressive symptoms and screen for depression among older people. It can be selfadministered or presented as an interview, and the questions have a yes/no format in order to be easy to understand for older people who may suffer from impaired cognitive function.
  This scale has 15 questions. In the assessment of the scale, no to positive questions and yes to negative questions were matched with 1 point and total score of 6 and above was considered significant for depressive symptoms.
Change in muscle strength | Baseline, 12th week
  The Jamar Handgrip Dynamometer is an instrument for measuring the maximum isometric strength of the hand and forearm muscles.
  The Takei Back and Leg Dynamometer measures peak pull force of the large muscle groups, these include: Legs,trunk,shoulders, arms.

CONTACTS AND LOCATIONS:
Overall Officials: Elvan Keleş, PT, PhD, Principal Investigator — İzmir Katip Çelebi Üniversitesi
Locations (1):
- Elvan Keleş, İzmi̇r, Turkey (Türkiye)